CLINICAL TRIAL: NCT01744613
Title: Clinical Impact of High on Treatment Platelet Reactivity Following Peripheral Endovascular Procedures. The PRECLOP Study (Platelet REsponsiveness to CLOpidogrel Treatment After Peripheral Angioplasty or Stenting)
Brief Title: High on Treatment Platelet Reactivity Following Peripheral Endovascular Procedures
Acronym: PRECLOP
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, SIABLIS DIMITRIOS, Dimitrios Siablis, Professor of Radiology, University of Patras
Other Study IDs: 822
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Influence of PRU Values on Primary Outcome
Keywords: Clopidogrel; platelet inhibition; antiplatelet therapy; peripheral arterial disease; endovascular treatment; angioplasty; stenting
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Will include patients with PRU values above the optimal cut-off value determined by ROC analysis
- Group B: Will include patients with PRU values below the optimal cut-off value determined by ROC analysis.

SUMMARY:
Antiplatelet therapy with clopidogrel is recommended following peripheral endovascular procedures. The clinical significance of an inadequate response to clopidogrel following percutaneous coronary interventions has been recently recognized.This study was designed to investigate platelet responsiveness to Clopidogrel following endovascular therapy of peripheral arterial disease using the VerifyNow P2Y12 point-of-care testing and to determine the optimal P2Y12 reactive unites (PRU) cut-off value of platelet inhibition influencing outcomes of infrainguinal angioplasty or stenting in patients receiving clopidogrel antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Rutherford 3-6 stage of peripheral arterial disease scheduled to undergo femoropopliteal or and infrapopliteal angioplasty or stenting.
* Patients receiving Clopidogrel per os 75 mg daily at least 1 month prior and 1 year after the procedure.

Exclusion Criteria:

* Acute limb ischemia
* Coagulation disorders
* Known allergy to clopidogrel
* Failure to comply with the antiplatelet treatment protocol
* Aortoiliac disease

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patient sampling of all patients undergoing pre-scheduled infrainguinal angioplasty or stenting due to symptomatic arterial disease in our Department from January 2010, treated with clopidogrel 75 mg daily.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Major event-free survival | 12 months
  12 months freedom from all causes of death, stroke, index limb amputation, non pre-scheduled minor amputation, index limb bypass surgery and target vessel recanalization (TVR)stratified according to PRU values distribution
Optimal P2Y12 reactive unites (PRU) cut-off value of platelet inhibition | 12 months
  Optimal P2Y12 reactive unites (PRU) cut-off value of platelet inhibition measured with VerifyNow P2Y12 assay point-of-care testing, influencing the 12 months primary outcome of major event-free survival estimated by ROC analysis

SECONDARY OUTCOMES:
Positive and negative predictive value of PRU testing | 12 months
  Positive and negative predictive value of PRU measurement with regard to the primary outcome of major event-free survival
Bleeding rate | 12 months
  12-months bleeding rate including intracranial hemorrhage and puncture related pseudoaneurysm stratified according to PRU values

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Siablis, MD, PhD, Study Director — University Hospital of Patras; Dimitrios Karnabatidis, MD, PhD, Principal Investigator — University Hospital of Patras; Stavros Spiliopoulos, MD, PhD, Principal Investigator — University Hospital of Patras; Georgios Pastromas, MD, Principal Investigator — University Hospital of Patras; Konstantinos Katsanos, MD, PhD, Principal Investigator — University Hospital of Patras
Locations (1):
- Patras University Hospital, Rio, Achaia, Greece

REFERENCES:
- [Derived] Spiliopoulos S, Pastromas G, Katsanos K, Kitrou P, Karnabatidis D, Siablis D. Platelet responsiveness to clopidogrel treatment after peripheral endovascular procedures: the PRECLOP study: clinical impact and optimal cutoff value of on-treatment high platelet reactivity. J Am Coll Cardiol. 2013 Jun 18;61(24):2428-2434. doi: 10.1016/j.jacc.2013.03.036. Epub 2013 Apr 16. PMID 23602777